CLINICAL TRIAL: NCT02814773
Title: Evaluation of the Quality of Life in the Elderly With Dementia : Validation of a Specific Instrument
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 112N04
Record Dates: First submitted 2016-06-16; First posted 2016-06-28 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- AD group: group suffering from Alzheimer-type dementia (mild to moderate dementia)
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires

SUMMARY:
With nearly one million cases of dementia in France in 2010, Alzheimer's disease (AD) and related syndromes are a major public health issue. The lake of drug for treatment or preventing AD, health related quality of life (HRQoL) became an essential criterion of evaluation to assess the treatment strategies of patients. Generic HRQoL tools are generally less sensitive for a given disease. That is why other specific tools for AD have been developed. None of them was validated in French. The aim of this study was therefore, after a review of the literature, to achieve a cross-cultural adaptation and psychometric validation of the "Quality of Life in Alzheimer's Disease" (QoL-AD) and "Dementia Quality of Life" (DQoL). These two questionnaires were selected because they were the most popular in English- language literature for this disease.This study concerned a total of 155 patient-caregiver pairs recruited from six French hospitals and a Francophone Swiss center. Patients had a confirmed diagnosis of AD (mild stage to moderate: Mini Mental State Examination ≥ 10). QoL-AD and DQoL were administered by an interviewer. The caregiver sheet of QoL-AD was self-administered. Cross-cultural adaptation and psychometric validation have been carried out for these two questionnaires.

DETAILED DESCRIPTION:
With nearly one million cases of dementia in France in 2010, Alzheimer's disease (AD) and related syndromes are a major public health issue. The lake of drug for treatment or preventing AD, health related quality of life (HRQoL) became an essential criterion of evaluation to assess the treatment strategies of patients. Generic HRQoL tools are generally less sensitive for a given disease. That is why other specific tools for AD have been developed. None of them was validated in French. The aim of this study was therefore, after a review of the literature, to achieve a cross-cultural adaptation and psychometric validation of the "Quality of Life in Alzheimer's Disease" (QoL-AD) and "Dementia Quality of Life" (DQoL). These two questionnaires were selected because they were the most popular in English- language literature for this disease.This study concerned a total of 155 patient-caregiver pairs recruited from six French hospitals and a Francophone Swiss center.

Patients had a confirmed diagnosis of AD (mild stage to moderate: Mini Mental State Examination ≥ 10). QoL-AD and DQoL were administered by an interviewer. The caregiver sheet of QoL-AD was self-administered. Cross-cultural adaptation and psychometric validation have been carried out for these two questionnaires. First step: the linguistic adaptation will be performed according to the latest available methodology: that of the " Institute for Work and Health ", as recommended 6 phases. Second step: the psychometric validation will be done after a multicentric study, cross repeated at weekly intervals for the validation phase , with two longitudinal points for the assessment phase of sensitivity to change. Analysis of the results will help define the applicability criteria and psychometric acceptability to know the validity of the adapted instrument that is to say, its content validity , validity of perceived, validity of structure, validity of agreement , its discriminative ability , reliability explored by internal consistency and stability over time. Longitudinal follow-up of patients is expected to also assess the sensitivity to change .

ELIGIBILITY:
To be included in the study, patients had to be :

* 65 years or older;
* native French speakers;
* living at home or in an institution;
* suffering from Alzheimer-type dementia defined according to DSM IV criteria, and had to obtain a score of 10 on the MMSE corresponding from mild to moderate dementia
* to have a main caregiver able to read.

Were not included in the cohort study , patients :

* From age 65;
* Achieved an evocative syndrome of dementia is not in accordance with the criteria DSM IV;
* From a mother tongue other than French;
* Possessing no help;
* With a MMSE score <10 , so with severe dementia;
* Hospitalized in short , medium or long stay;
* Having refused to participate in the study .

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients included were recruited in centres with a memory clinic or a geriatric ward.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2006-05; Primary Completion 2008-11 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The psychometric properties of QoL-AD and DQoL measured by questionnaire | 30 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, France, Reims, France

REFERENCES:
- [Result] Wolak A, Novella JA, Drame M, Morrone I, Boyer F, Blanchard F, Jolly D. Is the screening test of the French version of the dementia quality of life questionnaire indispensable? Dement Geriatr Cogn Dis Extra. 2011 Jan;1(1):84-92. doi: 10.1159/000326782. Epub 2011 Apr 6. PMID 22279447
- [Result] Wolak A, Novella JL, Drame M, Guillemin F, Di Pollina L, Ankri J, Aquino JP, Morrone I, Blanchard F, Jolly D. Transcultural adaptation and psychometric validation of a French-language version of the QoL-AD. Aging Ment Health. 2009 Jul;13(4):593-600. doi: 10.1080/13607860902774386. PMID 19629785
- [Result] Barbe C, Morrone I, Wolak-Thierry A, Drame M, Jolly D, Novella JL, Mahmoudi R. Impact of functional alterations on quality of life in patients with Alzheimer's disease. Aging Ment Health. 2017 May;21(5):571-576. doi: 10.1080/13607863.2015.1132674. Epub 2016 Jan 8. PMID 26745259
- [Derived] Barbe C, Jolly D, Morrone I, Wolak-Thierry A, Drame M, Novella JL, Mahmoudi R. Factors associated with quality of life in patients with Alzheimer's disease. BMC Geriatr. 2018 Jul 9;18(1):159. doi: 10.1186/s12877-018-0855-7. PMID 29986669